CLINICAL TRIAL: NCT01547338
Title: Comparison of Static Photography and Real Time Digital Video in the Assessment of Aesthetic Outcomes Following Breast Reconstruction
Brief Title: Photography or Video in Assessing Breast Reconstruction?
Status: Completed | Type: Observational
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Principal Investigator, Adam Gilmour, Clinical Laser Research Fellow, NHS Greater Glasgow and Clyde
Other Study IDs: GN12SU052
Record Dates: First submitted 2012-02-27; First posted 2012-03-07 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Breast Neoplasms; Breast Reconstruction
Keywords: Breast; Reconstruction
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Breast reconstruction patient: Unilateral breast reconstruction patients

SUMMARY:
Current qualitative methods of assessing the aesthetic result following breast reconstruction are known to be poor.

The investigators believe that real time digital video footage followed by expert panel review would be a superior method of qualitative assessment of breast cancer reconstruction aesthetics. This has never been studied before.

DETAILED DESCRIPTION:
Breast cancer is the commonest cancer to affect women in the UK. Current guidelines state that; disease permitting, all females due to undergo mastectomy for breast cancer should be offered reconstruction. This usually takes place in the form of implant based reconstruction, regional flap based reconstruction +/- implant or free autologous tissue based reconstruction.

Traditional methods of subjectively assessing the aesthetic outcome of any of the forms of breast surgery have been shown to be poor and the assessment of immediate reconstructions a cumbersome task. The qualitative part of the assessment usually relies on standardised clinical photographs and panel ratings. Four to six photographs are usually taken of the patient and their reconstruction from different angles. These photographs are then shown to an expert panel (usually consisting of healthcare professionals familiar with breast reconstruction).

A large degree of both inter and intra-observer bias exists when comparing standardized photographs. The results from expert assessment of cosmesis often do not correlate to the patients opinion with regards to the cosmetic outcome of their reconstruction

Due to the static nature of clinical photography it does not capture the effect which movement and gravity play on a reconstructed breast in comparison to a normal breast.

A large volume of information can be captured from a short digital video clip in comparison to a single photograph. The potential advantages of digital video assessment over photography are only beginning to be explored with regards to aesthetics in other fields associated to medicine.9 However this has never been trialed with regards to breast cancer reconstruction.

We believe that real time digital video footage would be a more valuable tool in the assessment of breast reconstruction. We believe that there may be more accurate correlations between patient's satisfaction and panel opinion and that there will be less inter and intra-observer discordance

ELIGIBILITY:
Inclusion Criteria:

* Female patient
* Minimum 18 years of age
* Due to attend for Nipple areola complex tattooing
* Previous unilateral breast reconstruction following mastectomy

Exclusion Criteria:

* Male patient
* Bilateral Breast Reconstruction
* Reconstruction less than 1year ago
* Breast reconstruction not following breast cancer excision

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast reconstruction patients attending for Nipple Areola Complex Tattoing
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2012-06; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Inter/Intra observer correlation on cosmetic scale using digital video footage | Outcome measure will be assessed approximately 1 year post breast reconstruction
  The primary aim of this study is to assess the level of inter and intra rater agreement for the expert panel on each of the 6 questions on the cosmetic outcome of breast reconstruction patients using digital video footage

SECONDARY OUTCOMES:
Comparison of digital video footage panel scores against patient self-assessment scores | Outcome measure will be assessed approximately 1 year post breast reconstruction
  If the above primary and secondary objectives show that the intra-observer agreement is good, to compare the agreement between patients' self-assessment and expert panel assessment

CONTACTS AND LOCATIONS:
Overall Officials: Adam Gilmour, MBChB, MRCS(Ed), Principal Investigator — NHS Greater Glasgow & Clyde
Locations (1):
- Canniesburn Plastic Surgery Unit, Glasgow Royal Infirmary, Glasgow, United Kingdom

REFERENCES:
- [Result] Gilmour A, Mackay IR, Young D, Hill ME, Brown L, Malyon AD. The use of real-time digital video in the assessment of post-operative outcomes of breast reconstruction. J Plast Reconstr Aesthet Surg. 2014 Oct;67(10):1357-63. doi: 10.1016/j.bjps.2014.05.036. Epub 2014 Jun 2. PMID 24923524